CLINICAL TRIAL: NCT05534360
Title: Tenecteplase Treatment in Ischemic Stroke Registry
Acronym: TETRIS
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220465
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Stroke, Acute
Keywords: Stroke; Ischemic stroke; Thrombolytic therapy; Tenecteplase; Thrombectomy; Cerebrovascular Disorders; Brain diseases; Central Nervous Diseases; Nervous system Diseases; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebrovascular Disorders; Brain Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tenecteplase: All consecutive patients with an arterial acute ischemic stroke treated with intravenous thrombolysis with tenecteplase.

SUMMARY:
The Tenecteplase Treatment in Acute Ischemic Stroke (TETRIS) Registry is multicenter ambispective observational study of patients with acute ischemic stroke who received intravenous thrombolysis with Tenecteplase

DETAILED DESCRIPTION:
Acute ischemic stroke management has considerably evolved over the last 20 years with the development of reperfusion treatments: intravenous thrombolysis (IVT) with alteplase, which is effective for AIS within 4.5 hours from symptoms onset and up to 9 hours in some cases; and mechanical thrombectomy (MT), in AIS with large vessel occlusion (LVO) within 24 hours from symptoms onset, either after IVT (bridging therapy) or alone in case of IVT contra-indication.

Alteplase is a recombinant form of tissue plasminogen activator (rtPA) that, when bound to fibrin, will activate plasminogen and lead to fibrinolysis and clot dissolution. It is administered at a dose of 0.9 mg/kg (maximum 90 mg) with an intravenous bolus (10% of the dose) followed by a one-hour infusion. Tenecteplase is a genetically modified form of alteplase with greater fibrin specificity and a longer half-life, which allows a simpler one bolus administration at a dose of 0.25 mg/kg (maximum 25 mg).

In the Tenecteplase versus Alteplase before Endovascular Therapy for Ischemic Stroke (EXTEND-IA TNK) randomized clinical trial, which compared tenecteplase and alteplase in bridging therapy for AIS with LVO, tenecteplase achieved a better recanalization rate on arteriography before MT and a better functional outcome at 3 months. Following this trial, tenecteplase was added in stroke guidelines as an alternative to alteplase for IVT in bridging therapy. More recently, the Alteplase compared to Tenecteplase (ACT) trial has shown, in patients with LVO and non-LVO AIS, that tenecteplase is non-inferior to alteplase in terms of functional outcome. It is likely that in the near future tenecteplase will be added as an alternative to alteplase for AIS without LVO. However, while some "real-life" studies have been published on tenecteplase use for AIS with LVO, data on the general use of tenecteplase are still scarce.

The Tenecteplase Treatment in Acute Ischemic Stroke (TETRIS) Registry is multicenter ambispective observational study of patients with acute ischemic stroke who received intravenous thrombolysis with Tenecteplase. The main aim of this registry is to provide routine clinical care data on the use of tenecteplase for IVT for both AIS with and without LVO, in order to further characterize the safety and efficacy of tenecteplase for AIS. Additionally, we aim to use this registry which combines clinical and radiological data to explore other aspects related to AIS management in this cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Confirmed acute arterial ischemic stroke on brain imaging (CT or MRI) within 270 minutes of symptoms onset or with perfusion CT or MRI criteria for an extended treatment window or wake-up strokes.
* Intravenous thrombolysis with tenecteplase

Exclusion Criteria:

* Contra-indication to intravenous thrombolysis
* Intravenous thrombolysis with alteplase
* Venous ischemic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients with an acute arterial ischemic stroke who received intravenous thrombolysis with tenecteplase in the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | Day 90
  Modified Rankin score (mRS), score ranging from 0 (no symptom) to 6 (death).

SECONDARY OUTCOMES:
Efficacy on functional independence (mRS ≤ 2) | Day 90
  Rate of functional independence defined as a modified Rankin score 0-2
Mortality rate | Day 90
  Rate of all-cause mortality
Early neurological outcome | Day 1
  National Institutes of Health Stroke Scale (NIHSS) score after 24 hours, ranging from 0 (no symptom) to 42 (death)
Incidence of haemorrhagic transformation | Day 1
  Incidence of intracerebral haemorrhage on MRI or CT after 24 hours (±12 hours) according to the ECASS II classification.
Incidence of symptomatic intracerebral haemorrhage (sICH) | Day 1
  Incidence of sICH according to the SITS-MOST definition.
Pre-thrombectomy recanalization rate | Day 1
  Rate of complete or near complete recanalization, defined as an extended Thrombolysis in Cerebral Infarction (mTICI) 2b50/2b66/2c/3 before thrombectomy
Final recanalization rate | Day 1
  Rate of complete or near complete recanalization after
Thrombolysis complication rate | Day 1
  Rate of complications linked to intravenous thrombolysis with tenecteplase
Thrombectomy complication rate | Day 1
  Rate of patients with secondary decompressive craniectomy

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Alamowitch, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Gaspard Gerschenfeld, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service des Urgences Cérébro-Vasculaires, Hôpitaux Universitaires Pitié-Salpêtrière et Saint-Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gerschenfeld G, Turc G, Obadia M, Chausson N, Consoli A, Olindo S, Caroff J, Marnat G, Blanc R, Ben Hassen W, Seners P, Guillon B, Wiener E, Bourcier R, Yger M, Cho TH, Checkouri T, Gory B, Smadja D, Sibon I, Richard S, Piotin M, Eker OF, Pico F, Lapergue B, Alamowitch S; for ETIS and TETRIS study groups. Functional Outcome and Hemorrhage Rates After Bridging Therapy With Tenecteplase or Alteplase in Patients With Large Ischemic Core. Neurology. 2024 Jul 9;103(1):e209398. doi: 10.1212/WNL.0000000000209398. Epub 2024 Jun 11. PMID 38862134
- See also: Institutional study link — https://institutducerveau-icm.org/fr/recherche-clinique/etudes-clinique/